CLINICAL TRIAL: NCT03014648
Title: A Phase II Clinical Trial Evaluating the Efficacy of Atezolizumab in Advanced Non-small Cell Lung Cancer (NSCLC) in Patients Previously Treated With PD-1-directed Therapy
Brief Title: Evaluating the Efficacy of Atezolizumab in Advanced Non-small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Liza Villaruz, MD (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Liza Villaruz, MD, Assistant Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC 16-153
Record Dates: First submitted 2016-12-29; First posted 2017-01-09 (Estimated); Results first posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-11

CONDITIONS: Advanced Non-small Cell Lung Cancer
MeSH Terms: interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Atezolizumab (Experimental): Atezolizumab will be given on day 1 of a 21-day cycle at 1200 mg IV over 60 (plus or minus 15) minutes for first infusion; can be decreased to 30 (plus or minus 10) minutes for subsequent cycles.
  Atezolizumab will be given as long as the patient continues to experience clinical benefit in the opinion of the investigator or until unacceptable toxicity, symptomatic deterioration attributed to disease progression.
  There will be no dose reduction for Atezolizumab. Patients may temporarily suspend study treatment for up to 84 days beyond the scheduled date of delayed infusion if study drug-related toxicity requiring dose suspension is experienced. If Atezolizumab is held because of adverse events for greater than 84 days beyond the scheduled date of infusion, the patient will be discontinued from Atezolizumab and will be followed for safety and efficacy.
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered through an IV over 60 minutes at a dose of 1200mg on Day 1 of each 21-day cycle. If the first dose is tolerated without any infusion-related adverse events, the following doses can be administered over 30 minutes.
  Other Names: Tecentriq

SUMMARY:
This is a phase II clinical trial aimed at evaluating the efficacy of PD-L1 inhibition with atezolizumab in advanced squamous and non-squamous NSCLC patients previously treated with anti-PD-1 therapy with either nivolumab or pembrolizumab.

In order to account for the variability of response kinetics to PD-1 directed therapy, patients will be enrolled in 3 parallel cohorts based on the best overall response to PD-1 directed therapy.

* Cohort 1 (progressive disease)
* Cohort 2 (stable disease with minimum 12 weeks of therapy)
* Cohort 3 (partial to complete response followed by progressive disease)

DETAILED DESCRIPTION:
Atezolizumab will be given on day 1 of a 21-day cycle at 1200 mg IV. Radiographic assessments for disease response will occur every 6 weeks while on treatment. Confirmatory scans should be obtained ≥ 4 weeks following initial documentation of objective response or progressive disease on atezolizumab therapy.

Atezolizumab will be given as long as the patient continues to experience clinical benefit in the opinion of the investigator or until unacceptable toxicity, symptomatic deterioration attributed to disease progression.

Patients will be followed for 12 months or until death as per standard of care after discontinuation of Atezolizumab or until death, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Stage IIIB/IV squamous or non-squamous NSCLC (American Joint Committee on Cancer 7th Edition Staging) who have had prior treatment with nivolumab or pembrolizumab will be enrolled in one of 3 parallel cohorts based on the following:

  * Cohort 1: Patient with progressive disease on nivolumab or pembrolizumab as the best overall response. Progressive disease must be confirmed with a confirmatory scan ≤ 4 weeks after the 1st documented date of progression.
  * Cohort 2: Patients with stable disease as the best overall response on a minimum of 12 weeks of therapy with nivolumab or pembrolizumab.
  * Cohort 3: Patients with partial or complete response as the best overall response followed by progressive disease, on nivolumab or pembrolizumab. A confirmatory scan at the time of disease progression must be performed ≤ 4 weeks after the 1st documented date of progression.
* Both men and women of all races and ethnic groups are eligible for this trial
* Patients must have resolution of toxic effects to Grade 1 or less from prior therapy (except alopecia).
* Patients must sign Informed Consent Form and show ability and willingness to comply with the requirements of the study protocol.
* 18 years of age or older
* Willingness to undergo a biopsy ≤ 6 weeks of the start of study treatment to obtain formalin-fixed paraffin-embedded tumor specimens in paraffin blocks (blocks are preferred) or at least 15 unstained slides, with an associated pathology report, for central testing of tumor PD-L1 expression.
* Adequate hematologic and end organ function, defined by the following laboratory results obtained within 14 days prior to the first study treatment (Cycle 1, Day 1):

  * ANC equal to/greater than 1500 cells/µL
  * WBC counts greater than 2500/µL
  * Lymphocyte count equal to/greater than 300µ/L
  * Platelet count equal to/greater than 100,000/µL
  * Hemoglobin equal to/greater than 9.0 g/dL
  * Total bilirubin equal to/less than 1.5 x ULN with the following exception:

    * Patients with known Gilbert disease who have serum bilirubin level equal to/less than 3 x ULN may be enrolled.
  * AST and ALT equal to/less than 3.0 x ULN with the following exception:

    * Patients with liver involvement: AST and/or ALT equal to/less than 5 x ULN
  * Alkaline phosphatase equal to/less than 2.5 x ULN with the following exception:

    * Patients with documented liver involvement or bone metastases: alkaline phosphatase equal to/less than 5 x ULN
* Serum creatinine equal to/less than 1.5 x ULN or creatinine clearance equal to/greater than 50 mL/min on the basis of the Cockcroft-Gault glomerular filtration rate estimation.
* Measurable disease per RECIST v1.1 for patients with solid malignancies.
* For female patients of childbearing potential and male patients with partners of childbearing potential, agreement (by patient and/or partner) to use highly effective form(s) of contraception (i.e., one that results in a low failure rate [less than 1% per year] when used consistently and correctly) and to continue its use for 5 months after the last dose of Atezolizumab.
* Eastern Cooperative Oncology Group Performance Status of 0 or 1. Patients with an ECOG Performance Status of 2 will be allowed at the discretion of the Treating Investigator in agreement with the Sponsor-Investigator.
* INR and aPTT equal to/less than 1.5 x ULN. This applies only to patients who do not receive therapeutic anticoagulation; patients receiving therapeutic anticoagulation (such as low-molecular-weight heparin or warfarin) should be on a stable dose.

Exclusion Criteria:

* Any approved anticancer therapy, including chemotherapy, hormonal therapy, or radiotherapy, within 3 weeks prior to initiation of study treatment; however, the following are allowed:

  * Hormone-replacement therapy or oral contraceptives.
  * Herbal therapy greater than 1 week prior to Cycle 1, Day 1 (herbal therapy intended as anticancer therapy must be discontinued at least 1 week prior to Cycle 1, Day 1).
  * Hormonal therapy for prostate cancer or breast cancer provided criteria in 3.2.21 are met.

    * Palliative radiotherapy (e.g., treatment of known bony metastases) allowed, provided it does not interfere with the assessment of tumor target lesions (e.g. the lesion being irradiated is not the only site of disease, because that would render the patient not evaluable for response by tumor assessments according to RECIST v1.1).
* Adverse events from prior anticancer therapy that have not resolved to Grade equal to/less than1 except for alopecia.
* History of grade 4 immune-related adverse events requiring treatment with prednisone or history of grade 3 immune-related adverse events requiring prednisone >10 mg/kg for >12 weeks.
* Bisphosphonate therapy for symptomatic hypercalcemia (use of bisphosphonate therapy for other reasons (e.g., bone metastasis or osteoporosis) is allowed).
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; cirrhosis; fatty liver; and inherited liver disease.
* Patients with acute leukemias, accelerated/blast phase chronic myelogenous leukemia, chronic lymphocytic leukemia, Burkitt lymphoma, plasma cell leukemia, or non-secretory myeloma.
* Known primary central nervous system (CNS) malignancy or symptomatic CNS metastases. Patients with asymptomatic untreated CNS disease may be enrolled, provided all of the following criteria are met:

  * Evaluable or measurable disease outside the CNS.
  * No metastases to brain stem, midbrain, pons, medulla, cerebellum, or within 10 mm of the optic apparatus (optic nerves and chiasm).
  * No history of intracranial hemorrhage or spinal cord hemorrhage.
  * No ongoing requirement for dexamethasone for CNS disease; patients on a stable dose of anticonvulsants are permitted.
  * No neurosurgical resection or brain biopsy within 28 days prior to Cycle 1, Day 1.
* Patients with asymptomatic treated CNS metastases may be enrolled, provided all the criteria listed above are met as well as the following:

  * Radiographic demonstration of improvement upon the completion of CNS directed therapy and no evidence of interim progression between the completion of CNS-directed therapy and the screening radiographic study.
  * No stereotactic radiation or whole-brain radiation within 28 days prior to Cycle 1, Day 1.
  * Screening CNS radiographic study equal to/greater than 4 weeks from completion of radiotherapy and equal to/greater than 2 weeks from discontinuation of corticosteroids.
* Patients who are pregnant, are lactation, or breastfeeding.
* Known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies.
* Inability to comply with study and follow-up procedures.
* History or risk of autoimmune disease, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Bell's palsy, Guillain-Barré syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis.

  * Patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone may be eligible.
  * Patients with controlled Type 1 diabetes mellitus on a stable insulin regimen may be eligible.
  * Patients with eczema, psoriasis, lichen simplex chronicus of vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:
  * Patients with psoriasis must have a baseline ophthalmologic exam to rule out ocular manifestations.
  * Rash must cover less than 10% of body surface area (BSA).
  * Disease is well controlled at baseline and only requiring low potency topical steroids (e.g., hydrocortisone 2.5%, hydrocortisone butyrate 0.1%, fluocinolone 0.01%, desonide 0.05%, alclometasone dipropionate 0.05%).
  * No acute exacerbations of underlying condition within the last 12 months (not requiring psoralen plus ultraviolet A radiation [PUVA], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors; high potency or oral steroids).
* History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest computed tomography (CT) scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications.
* History of HIV infection or active hepatitis B (chronic or acute) or hepatitis C infection.

  * Patients with past or resolved hepatitis B infection (defined as having a negative hepatitis B surface antigen [HBsAg] test and a positive anti-HBc [antibody to hepatitis B core antigen] antibody test) are eligible.
  * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
* Active tuberculosis.
* Severe infections within 4 weeks prior to Cycle 1, Day 1, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia.
* Signs or symptoms of infection within 2 weeks prior to Cycle 1, Day 1.
* Received oral or IV antibiotics within 2 weeks prior to Cycle 1, Day 1. Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible.
* Major surgical procedure within 28 days prior to Cycle 1, Day 1 or anticipation of need for a major surgical procedure during the course of the study.
* Administration of a live, attenuated vaccine within 4 weeks before enrollment or anticipation that such a live attenuated vaccine will be required during the study or for 5 months after the last dose of Atezolizumab. Influenza vaccination should be given during influenza season only (approximately October to March). Patients must not receive live, attenuated influenza vaccine (e.g., FluMist) within 4 weeks prior to enrollment, at any time during the study, or for 5 months after the last dose of Atezolizumab.
* Malignancies other than the disease under study within 5 years prior to Cycle 1, Day 1, with the exception of those with a negligible risk of metastasis or death and with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, or ductal carcinoma in situ treated surgically with curative intent) or undergoing active surveillance per standard-of-care management (e.g., chronic lymphocytic leukemia Rai Stage 0, prostate cancer with Gleason score equal to/less than 6, and prostate-specific antigen equal to/less than10 mg/mL, etc.).
* Treatment with investigational agent within 4 weeks prior to Cycle 1, Day 1 (or within five half lives of the investigational product, whichever is longer).
* Treatment with systemic immunosuppressive medications (including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to Cycle 1, Day 1.

  * Patients who have received acute, low dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled.
  * The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed.
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins.
* Patients with prior allogeneic bone marrow transplantation or prior solid organ transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Liza Villaruz, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (2):
- United States (2):
  - AdventHealth Orlando, Orlando, Florida
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Atezolizumab: Atezolizumab was administered through an IV over 60 minutes at a dose of 1200mg on Day 1 of each 21-day cycle. If the first dose was tolerated without any infusion-related adverse events, the following doses were administered over 30 minutes.
Period: Overall Study
Arm/Group | Atezolizumab
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients with advanced non-small cell lung cancer (NSCLC) patients previously treated with PD-1-directed therapy, treated with atezolizumab.
Groups:
- CR/PR Cohort: Patients with Complete Response (CR) or Partial Response (PR) Atezolizumab was given on Day 1 of a 21-day cycle at 1200 mg IV over 60 (plus or minus 15) minutes for first infusion, or decreased to 30 +/-10 min
- SD Cohort: Patients with Stable Disease (SD) Atezolizumab was given on Day 1 of a 21-day cycle at 1200 mg IV over 60 (plus or minus 15) minutes for first infusion, or decreased to 30 +/-10 min
- PD Cohort: Patients with Progressive Disease (PD) Atezolizumab was given on Day 1 of a 21-day cycle at 1200 mg IV over 60 (plus or minus 15) minutes for first infusion, or decreased to 30 +/-10 min
- Total: Total of all reporting groups
Arm/Group | CR/PR Cohort | SD Cohort | PD Cohort | Total
Number analyzed (Participants) | 8 | 3 | 17 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.50 (6.65) | 65.67 (13.65) | 66.41 (10.59) | 68.5 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 7 | 15
  Male | 3 | 0 | 10 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 2 | 2
  Unknown or Not Reported | 8 | 3 | 15 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 1 | 3
  White | 8 | 1 | 15 | 24
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Histology [Count of Participants; unit: Participants]
  ADENOCARCINOMA IN SITU, NOS | 0 | 0 | 1 | 1
  ADENOCARCINOMA, METASTATIC, NOS | 2 | 0 | 3 | 5
  ADENOCARCINOMA, N/A | 0 | 0 | 1 | 1
  ADENOCARCINOMA, NOS | 4 | 3 | 10 | 17
  LARGE CELL CARCINOMA, METASTATIC | 1 | 0 | 0 | 1
  NON-SMALL CELL CA | 0 | 0 | 1 | 1
  SQUAMOUS CELL CA METASTATIC, NOS | 0 | 0 | 1 | 1
  SQUAMOUS CELL CARCINOMA, NOS | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response (BOR)
Description: Best response recorded is recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started). Per RECIST v1.1: Complete Response (CR) - Disappearance of all target lesions. Any pathological lymph nodes (target or non-target) with reduction in short axis to <10 mm. Partial Response (PR): ≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Approximately 53.5 months
Population: Patients treated with atezolizumab who were previously treated with anti-PD-1 therapy and had at least one scan for evaluation of radiologic response.
Measure: Count of Participants; unit: Participants
Arm/Group | CR/PR Cohort | SD Cohort | PD Cohort
Number analyzed (Participants) | 7 | 3 | 16
Participants
  Progressive Disease | 2 | 2 | 9
  Partial Response | 1 | 0 | 1
  Stable Disease | 4 | 1 | 5
  Unknown | 0 | 0 | 1

2. Secondary Outcome: Duration of Response (DOR)
Description: The length of time that a tumor continues to respond to treatment from first documentation of response until disease progression.Per RECISIt v1.1: Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (target or non-target) with reduction in short axis to <10 mm. Partial Response (PR): ≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. Progressive Disease (PD):≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.
Time Frame: Approximately 56.5 months
Population: Patients treated with atezolizumab who were previously treated with anti-PD-1 therapy and evaluated for radiologic response.
Measure: Number; unit: months
Arm/Group | CR/PR Cohort | PD Cohort
Number analyzed (Participants) | 1 | 1
months | 6 | 0

3. Secondary Outcome: Progression-free Survival (PFS)
Description: The length of time during and after treatment that a patient lives with disease but without disease progression. Per RECISIT v1.1: Progressive Disease (PD):≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.
Time Frame: Approximately 56.5 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CR/PR Cohort | SD Cohort | PD Cohort
Number analyzed (Participants) | 8 | 3 | 17
months | 4.00 [2.00 to 9.00] | 2.00 [1.00 to NA] — Upper bound not reached | 2.00 [1.00 to 4.00]

4. Secondary Outcome: 6-month Progression-free Survival (PFS)
Description: The number of patients alive without disease progression at 6 months, per RECIST v1.1. Progressive Disease (PD):≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.
Time Frame: Up to 6 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | CR/PR Cohort | SD Cohort | PD Cohort
Number analyzed (Participants) | 8 | 3 | 17
Participants | 3 | 0 | 2

5. Secondary Outcome: 12-month Progression-free Survival (PFS)
Description: The number of patients alive without disease progression at 12 months, per RECIST v1.1. Progressive Disease (PD):≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.
Time Frame: Up to 12 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | CR/PR Cohort | SD Cohort | PD Cohort
Number analyzed (Participants) | 8 | 3 | 17
Participants | 1 | 0 | 1

6. Secondary Outcome: 24-month Progression-free Survival (PFS)
Description: The number of patients alive without disease progression at 24 months, per RECIST v1.1. Progressive Disease (PD):≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.
Time Frame: Up to 24 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- CR/PR Cohort: Patients with Complete Response (CR) or Partial Response(PR) Atezolizumab was given on Day1 of a 21-day cycle at 1200 mg IV over60 (plus or minus15) minutes for first infusion, or decreased to 30+/-10 min
Arm/Group | CR/PR Cohort | SD Cohort | PD Cohort
Number analyzed (Participants) | 8 | 3 | 17
Participants | 1 | 0 | 1

7. Secondary Outcome: Overall Survival (OS)
Description: The length of time from start of treatment that patients remain still alive.
Time Frame: Approximately 56.5 months
Population: All patients participating in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CR/PR Cohort | SD Cohort | PD Cohort
Number analyzed (Participants) | 8 | 3 | 17
months | 7.00 [2.00 to NA] — Upper 95% CI not reached | 11.00 [3.00 to NA] — Upper 95% CI not reached | 6.00 [4.00 to 11.00]

8. Secondary Outcome: 6-month Overall Survival (OS)
Description: The number of participants alive at 6 months.
Time Frame: Up to 6 months
Population: All study participants.
Measure: Count of Participants; unit: Participants
Arm/Group | CR/PR Cohort | SD Cohort | PD Cohort
Number analyzed (Participants) | 8 | 3 | 17
Participants | 4 | 2 | 8

9. Secondary Outcome: 12-month Overall Survival (OS)
Description: The number of patients alive at 12 months.
Time Frame: Up to 12 months
Population: All study participants.
Measure: Count of Participants; unit: Participants
Arm/Group | CR/PR Cohort | SD Cohort | PD Cohort
Number analyzed (Participants) | 8 | 3 | 17
Participants | 3 | 1 | 3

10. Secondary Outcome: 24-month Overall Survival (OS)
Description: The number of patients alive at 24 months.
Time Frame: Up to 24 months
Population: All study participants.
Measure: Count of Participants; unit: Participants
Arm/Group | CR/PR Cohort | SD Cohort | PD Cohort
Number analyzed (Participants) | 8 | 3 | 17
Participants | 1 | 0 | 1

11. Secondary Outcome: Adverse Events ≥ Grade 3
Description: Number of patients that experienced grade 3 or greater Adverse events per the Cancer Therapy Evaluation Program (CTEP) Common Terminology Criteria for Adverse Events (CTCAE) version 4, determined to be at least possibly, probably or definitely related to treatment, or that result in dose holds or reductions, will be collected and reported. Grade 3 = Severe AE and Grade 4 = Life-threatening or disabling AE. Adverse events and serious adverse events will be tabulated in order of prevalence, with the highest grade reported by each patient.
Time Frame: Approximately 56.5 months
Population: Patients treated with atezolizumab who were previously treated with anti-PD-1 therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | CR/PR Cohort | SD Cohort | PD Cohort
Number analyzed (Participants) | 8 | 3 | 17
Participants
  Diarrhea | 1 | 0 | 0
  Fatigue | 1 | 0 | 0
  Infusion related reaction | 1 | 0 | 0
  Lipase increased | 0 | 0 | 1
  Serum amylase increased | 0 | 0 | 1
  Generalized muscle weakness | 0 | 0 | 1

12. Other Pre Specified Outcome: PD-L1 Expression
Description: PD-L1 protein expression will be measured as positive (present) or negative (absent) in tissue from a biopsy conducted after discontinuation of the prior therapy and before initiation of study drug.
Time Frame: Up to 6 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Approximately 56.5 months
Description: CTCAE (4.0) Serious Adverse Events (SAE) are events ≥ Grade 3 Other Adverse Events (AE) are events ≤ Grade 2
Arm/Group | CR/PR Cohort | SD Cohort | PD Cohort
All-Cause Mortality (participants affected / at risk) | 8/8 | 3/3 | 17/17
Serious Adverse Events (participants affected / at risk) | 3/8 | 1/3 | 13/17
Other Adverse Events (participants affected / at risk) | 8/8 | 3/3 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CR/PR Cohort (N=8) | SD Cohort (N=3) | PD Cohort (N=17)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Asystole (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2
Colonic perforation (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 3
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2
Fever (General disorders) | 0 | 0 | 1
General disorders and administration site conditions - Other, specifyfailure to thrive (General disorders) | 0 | 0 | 1
Infusion related reaction (General disorders) | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 2
Specifycholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Abdominal infection (Infections and infestations) | 1 | 0 | 0
Lung infection (Infections and infestations) | 3 | 0 | 3
Sepsis (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Alkaline phosphatase increased (Investigations) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal and connective tissue disorder - Other, specifyRLE/R lower back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1
Paresthesia (Nervous system disorders) | 0 | 0 | 1
Stroke (Nervous system disorders) | 0 | 0 | 2
Confusion (Psychiatric disorders) | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CR/PR Cohort (N=8) | SD Cohort (N=3) | PD Cohort (N=17)
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 6 | 1 | 11
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Cardiac disorders - Other, specifyVolume overload (Cardiac disorders) | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 2
Sinus tachycardia (Cardiac disorders) | 4 | 1 | 3
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1
Endocrine disorders - Other, specifyTSH increase (Endocrine disorders) | 0 | 0 | 1
Endocrine disorders - Other, specifyTSH increased (Endocrine disorders) | 0 | 0 | 1
Endocrine disorders - Other, specifyelevated TSH (Endocrine disorders) | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 1
Glaucoma (Eye disorders) | 0 | 0 | 1
Blurred vision (Eye disorders) | 0 | 0 | 2
Esophagitis (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal disorders - Other, specifyhiatal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal disorders - Other, specifyloose stools (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 4
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 3
Diarrhea (Gastrointestinal disorders) | 2 | 0 | 5
Nausea (Gastrointestinal disorders) | 2 | 0 | 8
Constipation (Gastrointestinal disorders) | 3 | 0 | 5
Fever (General disorders) | 0 | 0 | 1
Localized edema (General disorders) | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 1
Neck edema (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1
Infusion related reaction (General disorders) | 0 | 1 | 0
Chills (General disorders) | 1 | 0 | 0
Edema limbs (General disorders) | 1 | 0 | 0
General disorders and administration site conditions - Other, specifypain, leg (General disorders) | 1 | 0 | 0
Flu like symptoms (General disorders) | 1 | 0 | 2
Fatigue (General disorders) | 4 | 1 | 9
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatobiliary disorders - Other, specifyLDH increased (Hepatobiliary disorders) | 1 | 0 | 0
Breast infection (Infections and infestations) | 0 | 0 | 1
Upper respiratory infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 3 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 2
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
INR increased (Investigations) | 0 | 0 | 1
Investigations - Other, specifyLDh increased (Investigations) | 0 | 0 | 1
Investigations - Other, specifyPT increased (Investigations) | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 2
Cardiac troponin T increased (Investigations) | 1 | 0 | 0
Hemoglobin increased (Investigations) | 1 | 0 | 0
Investigations - Other, specifythyroid stimulating hormone increased (Investigations) | 1 | 0 | 0
White blood cell decreased (Investigations) | 1 | 0 | 0
Creatinine increased (Investigations) | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 2
Lipase increased (Investigations) | 1 | 0 | 4
Alkaline phosphatase increased (Investigations) | 2 | 0 | 2
Investigations - Other, specifyLDH increased (Investigations) | 2 | 0 | 4
Serum amylase increased (Investigations) | 2 | 0 | 4
Weight loss (Investigations) | 3 | 0 | 1
Lymphocyte count decreased (Investigations) | 4 | 0 | 2
Activated partial thromboplastin time prolonged (Investigations) | 4 | 0 | 4
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0 | 3
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 4
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 4
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 0 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 0 | 4
Anorexia (Metabolism and nutrition disorders) | 4 | 0 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal and connective tissue disorder - Other, specifyBiopsy site pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal and connective tissue disorder - Other, specifyDJD - spine (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal and connective tissue disorder - Other, specifyL scapular pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal and connective tissue disorder - Other, specifyLL rib pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Dizziness (Nervous system disorders) | 0 | 0 | 2
Headache (Nervous system disorders) | 0 | 0 | 2
Paresthesia (Nervous system disorders) | 0 | 0 | 3
Confusion (Psychiatric disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 2
Agitation (Psychiatric disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Renal and urinary disorders - Other, specifyhesitancy (Renal and urinary disorders) | 0 | 0 | 1
Renal and urinary disorders - Other, specifymoderate bacteria in UA (Renal and urinary disorders) | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0
Urinary urgency (Renal and urinary disorders) | 1 | 0 | 0
Urine discoloration (Renal and urinary disorders) | 1 | 0 | 1
Hematuria (Renal and urinary disorders) | 1 | 0 | 2
Proteinuria (Renal and urinary disorders) | 2 | 0 | 4
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1
Scrotal pain (Reproductive system and breast disorders) | 0 | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, specifydecreased breath sounds (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, specifyhemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, specifyhemoptysis (intermittent) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, specifyupper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, specifyCOVID-19 (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, specifynonproductive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin and subcutaneous tissue disorders - Other, specifyBump in neck (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin and subcutaneous tissue disorders - Other, specifyL armpit lump (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin and subcutaneous tissue disorders - Other, specifyR lower breast (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin and subcutaneous tissue disorders - Other, specifyright forearm wound (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin and subcutaneous tissue disorders - Other, specifyskin tear on left arm (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Skin and subcutaneous tissue disorders - Other, specifyPruritus chest (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0
Hematoma (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 4
Hypotension (Vascular disorders) | 1 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-17): https://cdn.clinicaltrials.gov/large-docs/48/NCT03014648/Prot_SAP_000.pdf